CLINICAL TRIAL: NCT02595359
Title: Intracameral Moxifloxacin for Prevention of Postcataract Endophthalmitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Rodrigo Pessoa Cavalcanti Lira, Professor, Universidade Federal de Pernambuco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0001
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Endophthalmitis
Keywords: endophthalmitis; antibiotic therapy; cataract surgery; prevention
MeSH Terms: conditions — Endophthalmitis | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- moxifloxacin intracameral (Experimental): moxifloxacin injection given at conclusion of cataract intervention
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Moxifloxacin — Moxifloxacin intracameral
  Other Names: Vigamox

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of the prophylactic effect of intracameral moxifloxacin for prevention of postcataract endophthalmitis.

DETAILED DESCRIPTION:
Although cataract surgery is generally considered a safe procedure resulting in a favourable visual outcome, surgical complications do occur. The most feared complication is postoperative endophthalmitis which is an infectious condition caused by micro-organisms introduced to the interior of the eye during or after the surgical procedure.

As endophthalmitis is an infection, it should be preventable by antibiotic treatment.

Prophylactic antibiotic treatment can be given as topical treatment preoperatively, or during surgery directly into the anterior chamber, or as a subconjunctival, or it can be given as topical treatment postoperatively.

The aim of this study was to evaluate the efficacy and safety of the prophylactic effect of intracameral moxifloxacin for prevention of postcataract endophthalmitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of visually significant cataract

Exclusion Criteria:

* Has known allergies to moxifloxacin
* Has significant ocular co-morbidities in one or both eyes which may include (but is not limited to): advanced glaucoma, advanced or active macular degeneration, Fuchs corneal dystrophy, prior corneal transplantation, advanced diabetic eye disease, history of retinal detachment or any patient that would require billing a complex cataract procedure for any reason
* Has a known history of a condition which causes an immuno-compromised host state

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2013-01; Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
endothelial cell count | 6-month; 1 year; 2 years

SECONDARY OUTCOMES:
endophthalmitis incidence | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Lira, Principal Investigator — Prof
Locations (1):
- UFPE Ophthalmology, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
undecided